CLINICAL TRIAL: NCT00137241
Title: Determining the Prevalence of Health Literacy Among Veterans
Brief Title: Veterans as Leaders in Understanding and Education (VALUE)
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: CRI 03-153
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2006-10

CONDITIONS: Cancer
Keywords: health literacy; screening; cancer; health disparities
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1

SUMMARY:
The primary objectives for this study are to develop an estimate of the prevalence of health literacy at four geographically diverse Veterans Affairs Medical Centers (Minneapolis, Portland, Durham, and West Los Angeles), and for specific groups based on age, race, education, and geographic location. The investigators' secondary objectives are to illustrate the potential significance of poor health literacy by linking estimates for those over 50 years old to colorectal cancer (CRC) screening data and examining variation in screening rates by health literacy levels. The investigators expect that people with lower health literacy skills will be less adherent to CRC screening guidelines.

DETAILED DESCRIPTION:
BACKGROUND / RATIONALE:

Studies have shown that people with poor health literacy skills have significantly worse health status, greater risk for hospitalization, less knowledge about their health conditions, and are less likely to use preventative services. Little is known about the prevalence of low health literacy skills among veterans who use the VHA or the effect poor health literacy skills may have on complex preventative behaviors, such as screening for colorectal cancer (CRC). Understanding the distribution of health literacy skills among veterans and their effect on preventive behavior is critical for improving patient education, reducing health disparities, and promoting patient-centered care.

OBJECTIVE(S):

The primary objectives for this study are to develop an estimate of the prevalence of health literacy at four geographically diverse VAMCs (Minneapolis, Portland, Durham, and West LA), and for specific groups based on age, race, education, and geographic location. The secondary objectives are to link health literacy estimates for those 50 to 75 years old to CRC screening data, examine variation in guideline concordant screening rates by health literacy levels, and identify the mechanisms that may mediate or moderate the effect of health literacy on screening.

METHODS:

This observational study uses a time-sequential randomized design of 1440 veterans, stratified by age (<50, 50-75, >75), who have upcoming appointments in primary care clinics at the 4 study sites. Patients who are eligible (i.e., have at least 20/50 vision and are not demented) are asked to participate in a face-to-face structured survey with a study interviewer. The survey includes demographic data, functional status, social support, measures of attitudes and beliefs about health care providers, health insurers, medical care and the Short-Test of Functional Health Literacy in Adults (S-TOFHLA). For those between ages 50-75, knowledge of and attitudes towards CRC screening are also measured. Survey data are then matched to data from the CRC QUERI screening assessment and surveillance data system (CRS 02-162-1) to evaluate screening adherence.

STATUS:

Project work is ongoing.

IMPACT:

Findings from this study are expected to have a number of broad implications for research and practice within the VHA. This project will inform organizational changes aimed to improve the efficacy and efficiency of communication strategies and identify areas where interventions or system-level changes could be most effective; inform improvements in informed consent procedures, patient education, discharge summaries and prescription instructions; inform and improve the effectiveness of interventions and the Quality Enhancement and Research Initiative (QUERI) translation efforts; provide the basis for future longitudinal investigations into how health literacy changes over time; and, contribute to our understanding and amelioration of factors associated with health disparities.

ELIGIBILITY:
Inclusion Criteria:

All veterans eligible for care at any of the study facilities (Minneapolis, LA, Durham, and Portland VA Medical Centers) who were scheduled to have at least one primary care visit during the 6-month study recruitment period.

Exclusion Criteria:

Patients were excluded who had: 1) Severe cognitive disorders, 2) Severe visual impairment, 3) Severe hearing impairment, 4) Significant difficulty understanding English

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1850 (Estimated)
Dates: Start 2004-07; Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joan M. Griffin, PhD, Principal Investigator — Minneapolis VA Health Care System, Minneapolis, MN
Locations (1):
- Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota, United States

REFERENCES:
- [Result] Chew LD, Griffin JM, Partin MR, Noorbaloochi S, Grill JP, Snyder A, Bradley KA, Nugent SM, Baines AD, Vanryn M. Validation of screening questions for limited health literacy in a large VA outpatient population. J Gen Intern Med. 2008 May;23(5):561-6. doi: 10.1007/s11606-008-0520-5. Epub 2008 Mar 12. PMID 18335281
- [Result] Griffin JM, Partin MR, Noorbaloochi S, Grill JP, Saha S, Snyder A, Nugent S, Baines Simon A, Gralnek I, Provenzale D, van Ryn M. Variation in estimates of limited health literacy by assessment instruments and non-response bias. J Gen Intern Med. 2010 Jul;25(7):675-81. doi: 10.1007/s11606-010-1304-2. Epub 2010 Mar 12. PMID 20224964
- [Result] Griffin JM, Simon AB, Hulbert E, Stevenson J, Grill JP, Noorbaloochi S, Partin MR. A comparison of small monetary incentives to convert survey non-respondents: a randomized control trial. BMC Med Res Methodol. 2011 May 26;11:81. doi: 10.1186/1471-2288-11-81. PMID 21615955